CLINICAL TRIAL: NCT00303472
Title: An Open Label, Sequential Cohort, Dose Escalation Study to Evaluate the Safety and Efficacy of AMG 531 in Thrombocytopenic Subjects With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Brief Title: Determination of Safe Dose of Romiplostim (AMG 531) in Patients With Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050159; NCT00548028 (obsolete NCT alias)
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2010-11-19 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-11

CONDITIONS: Thrombocytopenia; MDS; Myelodysplastic Syndromes; Refractory Cytopenias
Keywords: MDS; Myelodysplastic Syndromes; Refractory Cytopenias; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia; Myelodysplastic Syndromes; Cytopenia | interventions — romiplostim

ARMS (7):
- Part A: 300 µg romiplostim (Experimental): Cohort 1 in Part A, participants received romiplostim 300 µg subcutaneously once weekly for 3 weeks. Participants who completed Part A could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
  Interventions: Drug: Romiplostim
- Part A: 700 µg romiplostim (Experimental): Cohort 2 in Part A, participants received romiplostim 700 µg subcutaneously once weekly for up to 3 weeks. Participants who completed Part A could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
  Interventions: Drug: Romiplostim
- Part A: 1000 µg romiplostim (Experimental): Cohort 3 in Part A, participants received romiplostim 1000 µg subcutaneously once weekly for up to 3 weeks. Participants who completed Part A could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
  Interventions: Drug: Romiplostim
- Part A: 1500 µg romiplostim (Experimental): Cohort 4 in Part A, participants received romiplostim 1500 µg subcutaneously once weekly for up to 3 weeks. Participants who completed Part A could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
  Interventions: Drug: Romiplostim
- Part B: 750 µg romiplostim SC QW (Experimental): Part B participants received romiplostim 750 µg subcutaneously (SC) once weekly (QW) for 8 weeks. Participants who complete Part B could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
  Interventions: Drug: Romiplostim
- Part B: 750 µg romiplostim SC Q2W (Experimental): Part B participants received romiplostim 750 µg subcutaneously every two weeks (Q2W) for 8 weeks. Participants who complete Part B could continue to receive injections of romiplostim for up to 1 year in the extension treatment phase.
  Interventions: Drug: Romiplostim
- Part B: 750 µg romiplostim IV Q2W (Experimental): Part B participants received romiplostim 750 µg intravenously (IV) once every two weeks for 8 weeks. Participants who complete Part B could continue to receive romiplostim for up to 1 year in the extension treatment phase.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim
  Other Names: AMG 531; Nplate®

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of romiplostim in thrombocytopenic patients with low or Intermediate-1 risk MDS. In addition, the study will evaluate the platelet response to romiplostim.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS using the World Health Organization classification
* Low or Intermediate-1 risk MDS using the International Prognostic Scoring System (IPSS)
* The mean of two platelet counts taken during the screening period must be ≤ 50 x 10^9/L, with no individual count > 55 x 10^9/L (The mean platelet counts of 5 subjects enrolled at the maximum tolerated dose (MTD) must be ≤ 20 x 10^9/L). Standard of care platelet assessments taken prior to Informed Consent may be used as 1 of the 2 counts taken within 3 weeks prior to study day 1.
* Must be ≥ 18 years of age at the time of obtaining informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at the time of screening
* Adequate Liver Function, as evidenced by a serum bilirubin ≤ 1.5 times the laboratory normal range (except for patients with a confirmed diagnosis of Gilbert's Disease), alanine aminotransferase (ALT) ≤ 3 times the laboratory normal range, and aspartate aminotransferase (AST) ≤ 3 times the laboratory normal range
* A serum creatinine concentration ≤ 2 mg/dL (≤ 176.6 µmol/L)
* Before any study-specific procedure, the appropriate written informed consent must be obtained (see Section 12.1)

Exclusion Criteria:

* Currently receiving any treatment for MDS other than transfusions and erythropoietic growth factors. If granulocyte growth factors are currently being received, they cannot be used on or after study day 1
* Clinically significant bleeding within 2 weeks prior to screening (eg, gastrointestinal (GI) bleeds, intracranial hemorrhage)
* Prior malignancy (other than controlled prostate cancer, in situ cervical cancer or basal cell cancer of the skin) unless treated with curative intent and without evidence of disease for ≥ 3 years before screening
* Prior history of bone marrow transplantation
* Persistent peripheral blood monocytosis (≥ 3 months with an absolute monocyte count > 1,000/µL)
* Unstable angina, congestive heart failure (New York Heart Association [NYHA] > class II), uncontrolled hypertension (diastolic > 100 mmHg), uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction
* Received Anti-Thymocyte Globuline (ATG) within 6 months of screening
* Received hypomethylating agents, immunomodulating agents, histone deacetylase inhibitors, cyclosporine or mycophenolate within 6 weeks of screening
* Received interleukin (IL)-11 (oprelvekin) within 4 weeks before screening
* Concurrent use of granulocyte growth factors (i.e. granulocyte-colony stimulating factor [G-CSF; Neupogen, Granocyte], pegfilgrastim [Neulasta], granulocyte macrophage-colony stimulating factor [GM-CSF; Leukine, Prokine, Sargramostim])
* Have ever previously received recombinant thrombopoietin (rTPO), pegylated recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF), eltrombopag, or romiplostim
* Less than 4 weeks since receipt of any therapeutic drug or device that is not Food and Drug Administration (FDA) approved for any indication
* Other investigational procedures are excluded
* History of arterial thrombosis (eg, stroke or transient ischemic attack) in the past year
* History of venous thrombosis that currently requires anti-coagulation therapy
* Untreated B12 or folate deficiency
* Subject is evidently pregnant (eg, positive human chorionic gonadotropin [HCG] test) or is breast feeding
* Subject is not using adequate contraceptive precautions
* Subject has known hypersensitivity to any recombinant E coli-derived product
* Subject previously has enrolled in this study
* Subject will not be available for follow-up assessment
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Kantarjian H, Fenaux P, Sekeres MA, Becker PS, Boruchov A, Bowen D, Hellstrom-Lindberg E, Larson RA, Lyons RM, Muus P, Shammo J, Siegel R, Hu K, Franklin J, Berger DP. Safety and efficacy of romiplostim in patients with lower-risk myelodysplastic syndrome and thrombocytopenia. J Clin Oncol. 2010 Jan 20;28(3):437-44. doi: 10.1200/JCO.2009.24.7999. Epub 2009 Dec 14. PMID 20008626
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 15-Feb-2006 Last Subject Enrolled: 29-Feb-2008
Pre-assignment Details: The study had 3 parts: Part A (4 weeks), Part B (8 weeks), and a treatment extension phase (up to 1 year). Subjects could participate in either Part A or Part B, and then could choose to enter the treatment extension phase. Subjects participating in Part A were not eligible for participation in Part B.
Groups:
- Part A: 300 µg Romiplostim: Cohort 1 in Part A participants received romiplostim 300 µg subcutaneously once weekly for 3 weeks. Participants who completed Part A could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
- Part B: 750 µg Romiplostim SC QW: Part B participants received romiplostim 750 µg subcutaneously (SC) once weekly (QW) for 8 weeks. Participants who completed Part B could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
- Part B: 750 µg Romiplostim SC Q2W: Part B participants received romiplostim 750 µg subcutaneously every two weeks (Q2W) for 8 weeks. Participants who completed Part B could continue to receive injections of romiplostim for up to 1 year in the extension treatment phase.
- Part B: 750 µg Romiplostim IV Q2W: Part B participants received romiplostim 750 µg intravenously (IV) once every two weeks for 8 weeks. Participants who completed Part B could continue to receive romiplostim for up to 1 year in the extension treatment phase.
Period: Treatment Period
Arm/Group | Part A: 300 µg Romiplostim | Part A: 700 µg Romiplostim | Part A: 1000 µg Romiplostim | Part A: 1500 µg Romiplostim | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Started | 6 | 11 | 11 | 16 | 11 | 12 | 5
Completed | 6 | 11 | 11 | 14 | 8 | 11 | 3
Not Completed | 0 | 0 | 0 | 2 | 3 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Disease Progression (to AML) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Extension (Optional)
Arm/Group | Part A: 300 µg Romiplostim | Part A: 700 µg Romiplostim | Part A: 1000 µg Romiplostim | Part A: 1500 µg Romiplostim | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Started | 6 | 11 | 11 | 13 | 5 | 5 | 1
Completed | 1 | 5 | 2 | 5 | 1 | 4 | 1
Not Completed | 5 | 6 | 9 | 8 | 4 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 4 | 2 | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2 | 1 | 0 | 0
Not completed — Other | 0 | 2 | 4 | 2 | 1 | 0 | 0
Not completed — Disease Progression (to AML) | 1 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: 300 µg Romiplostim: Cohort 1 in Part A, participants received romiplostim 300 µg subcutaneously once weekly for up to 3 weeks. Participants who completed Part A could continue to receive weekly injections of romiplostim for up to 1 year in the extension treatment phase.
- Total: Total of all reporting groups
Arm/Group | Part A: 300 µg Romiplostim | Part A: 700 µg Romiplostim | Part A: 1000 µg Romiplostim | Part A: 1500 µg Romiplostim | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W | Total
Number analyzed (Participants) | 6 | 11 | 11 | 16 | 11 | 12 | 5 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.5 (3.3) | 68.2 (10.2) | 70.9 (14.2) | 68.9 (13.8) | 69.4 (6.3) | 72.1 (9.9) | 72.2 (4.3) | 70.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 2 | 5 | 2 | 3 | 1 | 18
  Male | 6 | 6 | 9 | 11 | 9 | 9 | 4 | 54
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 5 | 11 | 9 | 14 | 10 | 10 | 4 | 63
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Japanese | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aborigine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Part A: Number of Participants With a Complete or Major Platelet Response
Description: Participants with a complete or major response during the treatment phase. A complete platelet response was defined as a platelet count ≥ 100 x 10^9/L during the treatment phase. A major platelet response was defined as an increase in absolute platelet count of ≥ 30 x 10^9/L for patients starting with > 20 x 10^9/L platelets, or an increase from ≤ 20 x 10^9/L to > 20 x 10^9/L and by at least 100%. Any participant receiving rescue medication was considered a non-responder. Platelet transfusions were considered rescue medication.
Time Frame: Treatment Period (4 weeks)
Population: Efficacy Analysis Set, composed of all enrolled participants who received romiplostim and completed the treatment phase.
Measure: Number; unit: Participants
Arm/Group | Part A: 300 µg Romiplostim | Part A: 700 µg Romiplostim | Part A: 1000 µg Romiplostim | Part A: 1500 µg Romiplostim
Number analyzed (Participants) | 6 | 11 | 11 | 16
Participants | 3 | 5 | 4 | 8

2. Secondary Outcome: Part B: Number of Participants With a Complete or Major Platelet Response
Description: as for outcome 1
Time Frame: Treatment Period (8 weeks)
Population: Efficacy Analysis Set, composed of all enrolled participants who received romiplostim and completed the treatment phase.
Measure: Number; unit: Participants
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 8 | 11 | 4
Participants | 5 | 8 | 2

3. Secondary Outcome: Part A: Number of Participants With a Platelet Response Per IWG Criteria
Description: The number of participants with a platelet response according to the modified International Working Group (IWG) criteria. Response was defined as an absolute increase of ≥ 30 x 10^9/L with Baseline platelet count > 20 x 10^9/L, or with a Baseline count ≤ 20 x 10^9/L, increasing to above 20 x 10^9/L and by at least 100% during the treatment or extension period and maintained for at least 8 consecutive weeks. Platelet transfusion was not considered a rescue medication but platelet counts ≤72 hours after platelet transfusion were excluded from the analysis.
Time Frame: Treatment period (4 weeks) and extension period (52 weeks).
Population: Subset of Efficacy Analysis Set, composed of all enrolled participants who received romiplostim and completed the treatment phase, who entered the treatment extension.
Measure: Number; unit: Participants
Arm/Group | Part A: 300 µg Romiplostim | Part A: 700 µg Romiplostim | Part A: 1000 µg Romiplostim | Part A: 1500 µg Romiplostim
Number analyzed (Participants) | 6 | 11 | 11 | 13
Participants | 3 | 6 | 4 | 6

4. Secondary Outcome: Part B: Number of Participants With a Platelet Response Per IWG
Description: as for outcome 3
Time Frame: Treatment period (8 weeks) and extension period (52 weeks).
Population: Efficacy Analysis Set, composed of all enrolled participants who received romiplostim and completed the treatment phase
Measure: Number; unit: Participants
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 8 | 11 | 4
Participants | 2 | 4 | 1

5. Secondary Outcome: Part B: Peak Platelet Count
Description: Peak platelet count (10^9/L) during the treatment period.
Time Frame: Treatment Period (8 weeks)
Population: Efficacy Analysis Set, composed of all enrolled participants who received romiplostim and completed the treatment phase.
Measure: Median (Inter-Quartile Range); unit: 10^9/L
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 8 | 11 | 4
10^9/L | 100.0 [49.0 to 175.5] | 111.0 [58.0 to 453.0] | 83.0 [55.0 to 135.0]

6. Secondary Outcome: Part B: Time to First Platelet Response
Description: Participants achieving first platelet response according to IWG criteria, by study week. Platelet response was defined as an absolute increase of ≥ 30 x 10^9/L with Baseline platelet count > 20 x 10^9/L, or with a Baseline ≤ 20 x 10^9/L increasing the platelet count to above 20 x 10^9/L and by at least 100% for 8 consecutive weeks. Platelet counts obtained within 72 hours of platelet transfusion were not evaluable for platelet response.
Time Frame: Treatment Period (8 weeks) and extension period (52 weeks).
Population: Efficacy Analysis Set, composed of all enrolled participants who received romiplostim and completed the treatment phase
Measure: Number; unit: Participants
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 8 | 11 | 4
Participants
  Week 1 Day 3 | 0 | 1 | 0
  Week 2 | 2 | 1 | 1
  Week 3 | 0 | 1 | 0
  Week 4 | 0 | 0 | 0
  Week 5 or later | 0 | 1 | 0
  Not Observed | 6 | 7 | 3

7. Secondary Outcome: Part B: Duration of Platelet Response
Description: Duration of platelet response per IWG criteria (absolute increase of ≥ 30 x 10^9/L with Baseline platelet count > 20 x 10^9/L, or with a Baseline ≤ 20 x 10^9/L increasing the platelet count to above 20 x 10^9/L and by at least 100% for 8 consecutive weeks).
Time Frame: Treatment Period (8 weeks) and extension period (52 weeks)
Population: Subset of Efficacy Analysis Set, composed of all enrolled participants who received romiplostim and completed the treatment phase, who had a platelet response
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 2 | 4 | 1
Weeks | 19.5 [8.0 to 31.0] | 9.0 [8.0 to 10.5] | 9.0 [9.0 to 9.0]

8. Secondary Outcome: Part B: Week 1 Cmax
Description: Maximum observed serum concentration (Cmax) of romiplostim during Week 1
Time Frame: Week 1
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 4 | 5 | 4
pg/mL | 3660 (3070) | 3190 (2360) | 197000 (112000)

9. Secondary Outcome: Part B: Week 1 Ctrough
Description: Measured romiplostim concentration at the end of the week 1 dosing interval (Ctrough)
Time Frame: Week 1
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 11 | 9 | 5
pg/mL | 171 (212) | 35.2 (31.5) | 96.5 (127)

10. Secondary Outcome: Part B: Week 1 AUC0-4
Description: Area under the romiplostim concentration-time curve from time zero to the last time point with quantifiable concentration (AUC0-4) during Week 1
Time Frame: Week 1
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 4 | 5 | 4
hr*pg/mL | 190000 (181000) | 182000 (111000) | 2030000 (838000)

11. Secondary Outcome: Part B: Week 7 Cmax
Description: Maximum observed serum concentration (Cmax) of romiplostim during Week 7.
Time Frame: Week 7
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W
Number analyzed (Participants) | 6 | 7
pg/mL | 785 (906) | 357 (361)

12. Secondary Outcome: Part B: Week 7 Ctrough
Description: Measured romiplostim concentration at the end of the Week 7 dosing interval (Ctrough)
Time Frame: Week 7
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W
Number analyzed (Participants) | 7 | 11
pg/mL | 54.6 (21.0) | 20.1 (1.98)

13. Secondary Outcome: Part B: Week 7 AUC0-4
Description: Area under the romiplostim concentration-time curve from time zero to the last time point with quantifiable concentration (AUC0-4) during Week 7.
Time Frame: Week 7
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W
Number analyzed (Participants) | 6 | 7
hr*pg/mL | 57100 (64300) | 35500 (36400)

14. Secondary Outcome: Part B: Week 1 Tmax
Description: Time at which the maximum concentration of romiplostum was observed after subcutaneous administration during Week 1
Time Frame: Week 1
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W
Number analyzed (Participants) | 4 | 5
Hours | 24.0 [24 to 24] | 24.0 [24 to 24]

15. Secondary Outcome: Part B: Week 7 Tmax
Description: Time at which the maximum concentration of romiplostum was observed after subcutaneous administration during Week 7
Time Frame: Week 7
Population: Safety Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W
Number analyzed (Participants) | 6 | 7
Hours | 24.0 [2 to 120] | 24.0 [24 to 72]

16. Primary Outcome: Part A: Number of Participants With Adverse Events
Description: The number of participants experiencing one or more adverse events during the treatment phase or extension phase of Part A.
Time Frame: Treatment period (4 weeks) plus treatment extension (1 year)
Population: All participants who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Part A: 300 µg Romiplostim | Part A: 700 µg Romiplostim | Part A: 1000 µg Romiplostim | Part A: 1500 µg Romiplostim
Number analyzed (Participants) | 6 | 11 | 11 | 16
Participants | 6 | 11 | 11 | 15

17. Primary Outcome: Part B: Number of Participants With Adverse Events
Description: The number of participants experiencing one or more adverse events during the treatment phase or extension phase of Part B.
Time Frame: Treatment period (8 weeks) plus treatment extension (1 year)
Population: All participants who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Number analyzed (Participants) | 11 | 12 | 5
Participants | 10 | 11 | 5

ADVERSE EVENTS:
Time Frame: Every visit and up to 30 days after end of study (up to 64 weeks)
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Part A: 300 µg Romiplostim | Part A: 700 µg Romiplostim | Part A: 1000 µg Romiplostim | Part A: 1500 µg Romiplostim | Part B: 750 µg Romiplostim SC QW | Part B: 750 µg Romiplostim SC Q2W | Part B: 750 µg Romiplostim IV Q2W
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/11 | 2/11 | 10/16 | 1/11 | 2/12 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 11/11 | 11/11 | 15/16 | 10/11 | 10/12 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 300 µg Romiplostim (N=6) | Part A: 700 µg Romiplostim (N=11) | Part A: 1000 µg Romiplostim (N=11) | Part A: 1500 µg Romiplostim (N=16) | Part B: 750 µg Romiplostim SC QW (N=11) | Part B: 750 µg Romiplostim SC Q2W (N=12) | Part B: 750 µg Romiplostim IV Q2W (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blast cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 300 µg Romiplostim (N=6) | Part A: 700 µg Romiplostim (N=11) | Part A: 1000 µg Romiplostim (N=11) | Part A: 1500 µg Romiplostim (N=16) | Part B: 750 µg Romiplostim SC QW (N=11) | Part B: 750 µg Romiplostim SC Q2W (N=12) | Part B: 750 µg Romiplostim IV Q2W (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lid lag (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scleritis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 5 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 5 | 2 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral mucosal petechiae (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 2 | 1 | 2 | 1 | 1
Catheter related complication (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 5 | 0 | 3 | 4 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 2 | 0 | 2 | 0 | 0
Infusion site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site haematoma (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 2 | 1 | 2 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 2 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 3 | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 2 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 1 | 4 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3 | 1 | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blast cell proliferation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 2 | 3 | 4 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bereavement reaction (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burnout syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 2 | 2 | 4 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.